CLINICAL TRIAL: NCT03597126
Title: Short Term Outcomes of Robotic-assisted Intersphincteric Resection for Low Rectal Cancer:A Multicentric Randomized Controlled Trial
Brief Title: Short Term Outcomes of Robotic-assisted Intersphincteric Resection for Low Rectal Cancer
Acronym: R-ISR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Li Chuan, Principal Investigator, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RoboticISR
Record Dates: First submitted 2018-04-23; First posted 2018-07-24 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Rectal Cancer
Keywords: Robotic; Intersphincteric Resection; rectal cancer; pelvic autonomic nerve anal function
MeSH Terms: conditions — Rectal Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot-assisted ISR (Active Comparator): Patients with low rectal cancer undergo intersphincteric resection assisted by Robotic
  Interventions: Device: Robot-assisted surgery
- laparoscopic ISR (Active Comparator): Patients with low rectal cancer undergo laparosocopic intersphincteric resection
  Interventions: Device: Laparoscopic surgery

INTERVENTIONS:
Device: Robot-assisted surgery — robot-assisted intersphincteric resection for low location rectal cancer(T=1&2)
  Arms: robot-assisted ISR
Device: Laparoscopic surgery — laparoscopic intersphincteric resection for low location rectal cancer(T=1&2)
  Arms: laparoscopic ISR

SUMMARY:
This study compared robot-assisted total mesorectal excision to treat very low rectal cancer within 2 cm from the dentate line to avoid permanent colostomy. improves the quality of life with better defecation function, urinary function and sexual function.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years < age < 80 years
2. Matching the diagnostic criteria;
3. tumor located 3 cm from anal verge
4. Clinically diagnosed cT1-3N0-2 M0 lesions
5. Tumor size of 4 cm or less
6. ASA 1-3 scores;
7. ECOG score is 0-1;
8. Adequate preoperative sphincter function

Exclusion Criteria:

1. Requiring a Mile's procedure
2. Fecal incontinence;
3. Previous abdominal surgery
4. Severe mental disease.
5. Intolerance of surgery for severe comorbidities
6. Emergency operation due to complication
7. Pregnant woman or lactating woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in urinary function | 6 months
  The days of indwelling catheter after operation The overall efficiency of urination function
Change in International Index of Erectile Function [IIEF] score | 18 months
  Alterations in IIEF scores from baseline up to 18 months postoperatively - 15 item questionnaire, each item range from 0 - 5, with total score to 30. lower score indicates more severe erectile dysfunction (ED)
Change in FIQL scores | 18 months
  Alterations in Fecal Incontinence Quality of Life Instrument (FIQL) scores from baseline up to 18 months postoperatively - 29 items range from 1 (strongly agree) to 4 (strongly disagree); with a 1 indicating a lower functional status of quality of life. Scale scores are only calculated if at least half of the items have been answered
Change in Female Sexual Function Index [FSFI] | 18 months
  Alterations in FSFI from baseline up to 18 months postoperatively - 19-item self-report measure, each item ranges from 0-5, with full range from 2 to 36, with low score indicating sexual function disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, China